CLINICAL TRIAL: NCT06245577
Title: Prospective Randomized Pilot Study on the Use of Biological Mesh Versus Synthetic Mesh in Interdisciplinary Resection Rectopexy With Sacro Colpopexy
Brief Title: Biological Mesh Versus Synthetic Mesh in Interdisciplinary RRP With SCP
Acronym: BioSynIRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelisches Klinikum Köln Weyertal gGmbH (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Principal Investigator, Claudia Rudroff, Consultant of the Deptartment of visceral surgery and functional surgery of the lower gastrointestinal tract, Evangelisches Klinikum Köln Weyertal gGmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EVKKoeln_BioSynIRS
Record Dates: First submitted 2024-01-18; First posted 2024-02-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Intestinal Obstruction; Pelvic Organ Prolapse; Rectal Prolapse
Keywords: rectopexy; sacro colpopexy
MeSH Terms: conditions — Intestinal Obstruction; Pelvic Organ Prolapse; Rectal Prolapse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: mesh material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomesh (Experimental): Biodesign (TM) Rectopexy Graft
  Mesh used in the mesh sacropexy of the middle pelvic organ compartment (vagina, cervix, or uterus); the mesh fixes the middle pelvic organ compartment to the promontory
  Interventions: Device: interdisciplinary mesh sacro colpopexy with resection rectopexy
- Synthetic mesh (Active Comparator): DynaMesh (TM) VASA
  Mesh used in the mesh sacropexy of the middle pelvic organ compartment (vagina, cervix, or uterus); the mesh fixes the middle pelvic organ compartment to the promontory
  Interventions: Device: interdisciplinary mesh sacro colpopexy with resection rectopexy

INTERVENTIONS:
Device: interdisciplinary mesh sacro colpopexy with resection rectopexy — surgical reconstruction of the middel pelvic compartment with the above mentioned meshes combined with a resection rectopexy in a simultaneous interdisciplinary procedure

SUMMARY:
The purpose of the pilot study is to demonstrate the safety and efficacy of a biological mesh compared to a standard synthetic mesh for the planned procedure in the above-mentioned clinical picture. Subsequently, a multicentre, randomized intervention study is planned to confirm the results and evaluate the long-term outcomes.

DETAILED DESCRIPTION:
Obstructive defecation syndrome (ODS) is a disordered defecation process due to a protrusion and telescope-like invagination of the lower rectum (rectocele, intussusception). This is often accompanied by a dolichocolon and chronic constipation. The feeling of an obstruction in the pelvic floor leads to forced pushing behavior in order to empty the rectum. Manual manipulation (transrectal or transvaginal) may also be necessary. Repeated and unsuccessful emptying attempts are often associated with the feeling of incomplete bowel evacuation. The patients affected are deeply frustrated and their thoughts revolve around the evacuation process. Their quality of life is considerably impaired. Around 10-25% of the population are affected The clinical picture predominantly affects women and is often associated with pelvic organ prolapse (POP). In these cases, the POP is the result of pathological pushing behavior for defecation. In addition, there may be other individual etiologies, such as post-vaginal delivery, connective tissue diseases, physiological lowering of the pelvic floor with age and surgical interventions in the pelvic area, which worsen the condition]. Up to 60% of the female population suffers from POP, and a third of these suffer from bowel dysfunction in the form of constipation (33%) and/or ODS (26%).

Conservative treatment options such as dietary changes, adequate fluid intake, laxative medication, physical exercise, pelvic floor training, pelvic floor biofeedback therapy with or without electro stimulation and pessary treatment are limited and do not achieve the desired long-term effect Surgery is the alternative in these cases with the aim of restoring the anatomy More than 12% of all women have to undergo surgery in the course of their lives For some time now, an interdisciplinary surgical approach has been possible in which all affected compartments can be treated in a single procedure. The current results demonstrate the safety of this approach and represent a promising option for affected patients.

At the same time, the US Food and Drug Administration (FDA) issued a warning in 2008 against the use of mesh implants in reconstructive pelvic floor surgery, as serious long-term complications have sometimes been observed. With synthetic mesh, the mesh remains permanently in close proximity to the other pelvic organs and can lead to mesh infection, erosion and migration over time. These conditions can have serious consequences for individual patients and in some cases even lead to a permanent stoma. The use of synthetic mesh is restricted in the United States for both transvaginal and abdominal POP surgery due to long-term complications (erosion, migration and chronic infection of the mesh). In Germany, the use of synthetic meshes is also highly controversial and is restricted to use in POP with vaginal reconstruction for recurrent procedures.

The information about serious adverse events associated with the use of synthetic mesh in reconstructive pelvic floor surgery has unsettled many patients. Women of a younger age in particular have a long life expectancy and an increased risk of adverse events due to the synthetic mesh material. Some of them still want to become pregnant after the operation. At the same time, the disease - even if it is not life-threatening - has an enormous impact on the individual's quality of life, and most of those affected still need surgery.

For these patients, the use of a biological mesh appears to be a sensible alternative. The biological material carries a low risk of mesh infection, as the material allows cellular infiltration and is degraded within 12 to 18 months. There is no risk of arrosion or migration of the biological mesh due to the degradation of the material. However, the reconstruction may lose its stability after degradation of the mesh, which in some cases could lead to recurrence of the depression. This in turn could reduce the long-term success of the intervention. This is possibly the reason why the biological mesh is currently not recommended for SCP in the German guideline for pelvic floor surgery . However, there is little scientific evidence and the recommendation in the guideline is based on only two publications on this topic. At the same time, biological meshes have been used for ventral mesh rectopexy for some time with promising results. No mesh-related complications have yet been observed. As a result, the Biodesign rectopexy graft received FDA approval in the USA and CE marking in Germany in accordance with the Medical Device Directive.

The data on the use of biological mesh for ventral mesh rectopexy and the wishes of the patients concerned have encouraged us to re-evaluate the issue. We are convinced that the bionet leads to the formation of scar tissue during apical fixation of the internal genitalia by means of sacrocolpopexy and in combination with resection rectopexy, which fixes the pelvic organs in place even after resorption of the mesh and prevents recurrence of descensus.

In the study, the mesh is placed in the same space (between the rectum and vagina) as for the treatment of rectal prolapse/intussusception in mesh rectopexy. With this defined and standardized technique, Cook Biotech evaluates the mesh application in this pilot study as "intended use" of its approved product. Furthermore, the Ethics Committee of the University of Cologne confirms that the biological mesh is used for this pilot study within the scope of its intended purpose and in accordance with the safety and quality requirements of the European Medical Device Regulation (MDR). Thus, the study falls under §47 (3) of the MDR.

The planned pilot study is necessary in view of the currently still negative recommendation of the German guideline, the limited data on the use of biological mesh in laparoscopic SCP and the risks associated with the use of synthetic mesh, especially in younger women, in order to find an alternative to the synthetic mesh material.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of obstructed defection syndrome
* clinical diagnosis of pelvic organ prolapse pelvic organ prolapse
* must be suitable for surgery

Exclusion Criteria:

* allergy to the components of the mesh
* pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
safety of the experimental internvention as measured by surgical outcome | 12 months
  Morbidity and mortality according to the Clavien-Dindo Classification (CDC) at 12 months after surgery (maximum value)

SECONDARY OUTCOMES:
Altomare Score for Obstruct4ed defecation syndrome (ODS) | 12 months
  Improvement in medical condition as measured Altomare score for ODS, min/max points 0-30 point, more points indicate more severe ODS symptoms; a reduction after intervention indicatesmprovement/deterioration (-3 =better, - 6 = much better; +3=worse, +6=much worse)
Pelvic organ prolapse Quantification (POP Q) | 12 months
  Measurement of clinical pelvic organ prolapse by the above score. min/max 0-4, more points are more symptoms. Improvement of the POP-Q is -1= good; -2 = very good; +1 =worse, +2=much worse.
Rectal Toxicity Score for bowel dysfunction | 12 months
  Improvement in medical condition as measured rectal toxicity score for bowel dysfunction, min/max points 0-30 point, more points indicate more severe bowel dysfunction; a reduction after intervention indicates improvement/deterioration (-3 =better, - 6 = much better; +3=worse, +6=much worse)
Wexner Incontinence Score for fecal incontinence | 12 months
  Improvement in medical condition as measured with Wexner Incontinence Score for fecal incontinence, min/max points 0-20 point, more points indicate more severe incontinence symptoms; a reduction after intervention indicates mprovement/deterioration (-3 =better, - 6 = much better; +3=worse, +6=much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Privatdozentin c Rudroff, Principal Investigator — Evagelisches Klinikum Koeln Weyerta
Locations (1):
- Evangelisches Klinikum Koeln Weyertal, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
no IPD will be available. The Study protocol and the informed consent form are available upon request. After closure of the study the de-identified participant data may be requested through the clinical principal investigator
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: are available and may be requested until closure of the trial
Access Criteria: request via email to the principal investigator

REFERENCES:
- [Background] Brunner M, Roth H, Gunther K, Grutzmann R, Matzel KE. Ventral rectopexy with biological mesh: short-term functional results. Int J Colorectal Dis. 2018 Apr;33(4):449-457. doi: 10.1007/s00384-018-2972-3. Epub 2018 Feb 13. PMID 29442156
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Augusto KL, Bezerra LRPS, Murad-Regadas SM, Vasconcelos Neto JA, Vasconcelos CTM, Karbage SAL, Bilhar APM, Regadas FSP. Defecatory dysfunction and fecal incontinence in women with or without posterior vaginal wall prolapse as measured by pelvic organ prolapse quantification (POP-Q). Eur J Obstet Gynecol Reprod Biol. 2017 Jul;214:50-55. doi: 10.1016/j.ejogrb.2017.04.039. Epub 2017 Apr 26. PMID 28477524
- [Background] Sohlberg EM, Dallas KB, Weeks BT, Elliott CS, Rogo-Gupta L. Reoperation rates for pelvic organ prolapse repairs with biologic and synthetic grafts in a large population-based cohort. Int Urogynecol J. 2020 Feb;31(2):291-301. doi: 10.1007/s00192-019-04035-3. Epub 2019 Jul 12. PMID 31312846
- [Background] Ahmad M, Sileri P, Franceschilli L, Mercer-Jones M. The role of biologics in pelvic floor surgery. Colorectal Dis. 2012 Dec;14 Suppl 3:19-23. doi: 10.1111/codi.12045. PMID 23136820
- [Background] de Mattos Lourenco TR, Pergialiotis V, Durnea C, Elfituri A, Haddad JM, Betschart C, Falconi G, Doumouchtsis SK; CHORUS: An International Collaboration for Harmonising Outcomes, Research, and Standards in Urogynaecology and Women's Health. A systematic review of reported outcomes and outcome measures in randomized controlled trials on apical prolapse surgery. Int J Gynaecol Obstet. 2019 Apr;145(1):4-11. doi: 10.1002/ijgo.12766. Epub 2019 Feb 22. PMID 30671950
- [Background] Clemons JL, Weinstein M, Guess MK, Alperin M, Moalli P, Gregory WT, Lukacz ES, Sung VW, Chen BH, Bradley CS; AUGS Research Committee. Impact of the 2011 FDA transvaginal mesh safety update on AUGS members' use of synthetic mesh and biologic grafts in pelvic reconstructive surgery. Female Pelvic Med Reconstr Surg. 2013 Jul-Aug;19(4):191-8. doi: 10.1097/SPV.0b013e31829099c1. PMID 23797515

DOCUMENTS (1):
  • Informed Consent Form (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT06245577/ICF_001.pdf